CLINICAL TRIAL: NCT00147069
Title: Investigation Into Inflammatory Mechanisms in Airway Cells in Smokers and Non-smokers With Inflammatory Lung Disease.
Brief Title: Leukocyte Function in Asthma and COPD
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 04-059
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Asthma; COPD; Emphysema; Chronic Bronchitis
Keywords: sputum; macrophage; neutrophil
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Controls: Non-smoking control subjects without lung disease
- Asthmatics: Non-smokers patients with asthma
- Non-COPD smokers: Current smokers without airways obstruction, FEV1 >80% predicted
- COPD smokers: Patients with COPD and cigarette smokers

SUMMARY:
The aim of this study is to examine the inflammatory mechanisms involved in the pathogenesis of inflammatory lung disease, in particular to compare the inflammatory profile seen in asthma and COPD. Evidence for inflammation in asthma and COPD is based on the finding of increased numbers of macrophages and neutrophils in the lungs and respiratory secretions of these patients. The inflammatory cells produce proteases, as well as, reactive oxidant species resulting in a protease/anti-protease imbalance which favours lung destruction. The aim is to examine the inflammatory mediators released by inflammatory cells (such as, macrophages and lymphocytes) in order to determine whether there are differences between non-smoking subjects, smoking subjects and patients with asthma or COPD. Monocytes are precursors of alveolar macrophages, and both monocytes and neutrophils are recruited to the lung from the blood via the action of specific chemoattractants. We have evidence that in inflammation there are higher levels of these chemoattractants. Therefore these cells might also demonstrate the same changes seen in alveolar macrophages from these patients.

We also aim to assess the role of the macrophage precursor (monocyte) and neutrophils in the blood. We will also assess lymphocyte/monocyte interaction. We will do this as the lymphocyte may be involved in the initial recruitment of inflammatory cells. We will also assess the role of cytokines involved with monocyte/macrophage/neutrophil migration in induced sputum as well as the role of induced sputum in the migration of monocytes and neutrophils into the lung. Our aim is to link the initial changes in blood to the changes causing disease in the lungs. We aim to examine cellular responses in four groups of subjects, namely (i) non-smoking controls, (ii) smokers without clinical evidence of COPD or asthma, (iii) smokers with COPD (iv) asthmatic patients.

DETAILED DESCRIPTION:
Overall subjects will be characterised into one of four groups: normal non-smoking subjects, healthy smokers, patients with asthma and patients with COPD. Subjects will have had to fulfil inclusion and exclusion criteria, and give written consent.

Recruitment Methods. Volunteer subjects (healthy non-smokers and healthy smokers) will be recruited from within the National Heart and Lung Institute. Volunteers will be recruited via advertising using ethically approved advertisements. Asthmatic and COPD patients will be recruited from the outpatient clinic at The Royal Brompton Hospital. At the screening visit, the diagnosis of asthma or COPD will be confirmed from the clinical case notes. If the patient is a volunteer, they will undergo a full history and examination, spirometry. Each subject will attend on one study visit only. At the first visit a number of investigations will be undertaken including, spirometry with reversibility (400 microg ventolin via metered dose inhaler if initial spirometry shows an obstructive picture to exclude asthmatics), and sputum induction. In addition, 50ml of venous blood will be taken.

More specifically, the following interventions will be undertaken by each subject

1. Medical History and Physical Examination A full medical history and physical examination (including height and weight) will be performed on the initial screening visit, in addition to that recorded in the clinical case notes.
2. Respiratory Assessments Forced Expiratory Volume per second (FEVI) will be measured using a dry wedge spirometer (Vitalograph, Buckingham, UK) and expressed as a percent of predicted value. Subjects will be trained in the use of the apparatus before beginning the study. The baseline value at each visit will be measured after at least fifteen minutes of quiet rest, and will be taken as the highest of three readings made at one minute intervals. 400 microg ventolin administered via a metered dose inhaler will be given if initial spirometry shows an obstructive picture (FEV1 <80% predicted, FEV1 /FVC<70%) in order to distinguish between the presence of asthma or COPD.
3. Sputum Induction Sputum induction will be performed in the Asthma Laboratory. The subject will inhale 3.5% saline at room temperature, nebulised via a De Vilbiss 99 Ultrasonic nebuliser set, at maximum output using a mouthpiece. After five minutes the subject will rinse his/her mouth thoroughly with water, and will be asked to cough deeply and expectorate sputum into a pot. Samples from this first five minute collection are discarded. This procedure will continue for a further ten minutes, and the resulting sample will be collected in a polypropylene pot.

   It is important to explain to the subject that the aim is to obtain sputum, and that saliva should be disposed of by spitting into a bowl which is later discarded.

   In the case of any chest discomfort or shortness of breath, the procedure is stopped and spirometry is repeated. If the FEV1 has fallen by 10% of the predicted value, the subject can rest until the FEV1 has returned to the baseline value or the procedure can be terminated.

   Sputum samples will be analysed for differential and absolute cell counts (eosinophils, neutrophils, macrophages, lymphocytes, and columnar epithelial cells). Sputum supernatants will be assayed for TNF-alpha, IL-8, interferon-gamma, and other cytokine levels.

   Immunohistochemistry will be performed on the induced sputum samples to identify the cellular localisation of factors involved with leukocyte function.

   Cytospin preparations will be made for differential cell counts and the soluble fraction will be used for cytokine assays.
4. Venous Blood Sampling Fifty (50) millilitres of blood shall be venesected at the study visit. We will investigate factors involved in leukocyte function and chemotaxis. We will also assess cellular distributions of receptors thought to be important in regulation by using FACS analysis.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic patients:

1. Age 21-79 years of both sexes (females will be taking adequate contraceptive measures).
2. Increase in FEV1 >15% and >200ml following beta2 agonist inhalation, either at the time of study or previously documented

COPD patients:

1. Stable patients with a post-salbutamol FEV1 30-70% predicted normal of >1L
2. Increase in FEV1 < 15% and < 200 ml following beta2 agonist inhalation, either at the time of study or previously documented
3. Age 21-79 years of both sexes (females will be taking adequate contraceptive measures )
4. Smokers
5. No history of allergic or respiratory disease.

Normal Volunteers

1. Age 21-79 years of both sexes (females will be taking adequate contraceptive measures )
2. Non-smokers
3. Normal lung function
4. No upper respiratory tract infection within the last 4 weeks
5. No history of allergic or respiratory disease.

Healthy Smokers 1. Age 21-79 years of both sexes (females will be taking adequate contraceptive measures ) 2. Smokers 3. Normal lung function 4. No upper respiratory tract infection within the last 4 weeks

-

Exclusion Criteria:

1. Asthmatic patients with FEV1 less than 40% predicted value
2. Alcohol abuse
3. Any history or evidence of hepatic, cardiovascular or renal disease
4. Any history or evidence of neuropsychiatric disease
5. Drug abuse or any other condition associated with poor compliance
6. Pregnancy or breast feeding
7. Patients are unable to provide written informed consent

COPD patients:

1. Any other active lung diseases 2. Upper respiratory infection within the last 4 weeks 3. Pregnancy or breast feeding 4. Any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study 5. Subjects unable to give informed consent

-

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four groups of subjects were recruited: patients with COPD (cigarette smokers), diagnosed according to current standard criteria, patients with asthma (non-smokers), diagnosed according to current standard criteria, including a personal history of asthma, current smokers without airways obstruction (FEV1480% predicted) and non-smoking control subjects without lung disease
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise E Donnelly, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital/NHLI Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Culpitt SV, Rogers DF, Traves SL, Barnes PJ, Donnelly LE. Sputum matrix metalloproteases: comparison between chronic obstructive pulmonary disease and asthma. Respir Med. 2005 Jun;99(6):703-10. doi: 10.1016/j.rmed.2004.10.022. Epub 2004 Dec 13. PMID 15878486

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Controls | Asthmatics | Non-COPD Smokers | COPD Smokers
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | Asthmatics | Non-COPD Smokers | COPD Smokers | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (1.4) | 34.6 (1.6) | 47.6 (2.6) | 60.7 (2.6) | 43.3 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 10 | 3 | 31
  Male | 6 | 6 | 5 | 12 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 15 | 15 | 15 | 60
FEV1 percent predicted [Mean (Standard Deviation); unit: percent predicted] | 104.9 (1.7) | 93.5 (1.1) | 100.9 (1.2) | 45.2 (3.1) | 86 (7)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Inflammatory Cells Recovered in Sputum
Description: Sputum was induced via inhalation of hypertonic saline as previously described, and was processed for differential counts of inflammatory cells.
Time Frame: 1 year
Measure: Mean (Standard Error); unit: 10^6 cells/ml
Arm/Group | Controls | Asthmatics | Non-COPD Smokers | COPD Smokers
Number analyzed (Participants) | 15 | 15 | 15 | 15
10^6 cells/ml | 2.3 (0.5) | 2.1 (0.4) | 1.9 (0.3) | 5.2 (1.5)
Statistical Analysis 1: Comparison: Controls vs Asthmatics vs Non-COPD Smokers vs COPD Smokers; Test type: Superiority; p = 0.1, Kruskal-Wallis

2. Primary Outcome: Number of Matrix Metalloproteases (MMPs) MMP1
Description: MMPs determined using paired antibody quantitative ELISAs
Time Frame: 1 year
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Controls | Asthmatics | Non-COPD Smokers | COPD Smokers
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng/ml | 11.0 (1.5) | 12.5 (1.7) | 16.5 (0.6) | 34.5 (3.2)
Statistical Analysis 1: Comparison: Controls vs Asthmatics vs Non-COPD Smokers vs COPD Smokers; Test type: Superiority; p = 0.05, Kruskal-Wallis — The reported p value was calculated

3. Primary Outcome: Number of Matrix Metalloproteases (MMPs) MMP3
Description: MMPs determined using paired antibody quantitative ELISAs
Time Frame: 1 year
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Controls | Asthmatics | Non-COPD Smokers | COPD Smokers
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng/ml | 7.2 (1.4) | 4.5 (0.8) | 5.8 (1.7) | 5.4 (1.1)
Statistical Analysis 1: Comparison: Controls vs Asthmatics vs Non-COPD Smokers vs COPD Smokers; Test type: Superiority; p = 0.05, Kruskal-Wallis

4. Primary Outcome: Number of Matrix Metalloproteases (MMPs) MMP8
Description: MMPs determined using paired antibody quantitative ELISAs
Time Frame: 1 year
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Controls | Asthmatics | Non-COPD Smokers | COPD Smokers
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng/ml | 208.6 (24.7) | 188.5 (29.4) | 443.5 (72) | 1575 (521)
Statistical Analysis 1: Comparison: Controls vs Asthmatics vs Non-COPD Smokers vs COPD Smokers; Test type: Superiority; p = 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Controls | Asthmatics | Non-COPD Smokers | COPD Smokers
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes